CLINICAL TRIAL: NCT01207180
Title: Discharge Planning for Elderly Patients in the Emergency Department: Use of a Brief Phone Call After Discharge to Improve Medication Utilization and Physician Follow-up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: The Duke Endowment (Other)
Responsible Party: Principal Investigator, Kevin Biese, MD, Assistant Professor of Emergency Medicine, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 10-0978
Record Dates: First submitted 2010-09-13; First posted 2010-09-22 (Estimated); Last update posted 2011-11-18 (Estimated); Status verified 2011-11

CONDITIONS: Patient Discharge
Keywords: emergency medicine; primary care physicians

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Follow-up phone call from Nurse (Experimental): Patients in this are will receive a phone call follow-up from a nurse 1-3 days after their discharge from the ED.
  Interventions: Other: Phone call follow-up
- Satisfaction survey (Placebo Comparator): This group of patients will receive a phone call from a student who will conduct a brief satisfaction survey of the patient's experience in the ED.
  Interventions: Other: Satisfaction survey
- Control group (Placebo Comparator): Patients in this group will receive no phone call at 1-3 days.
  Interventions: Other: Control group --- no intervention

INTERVENTIONS:
Other: Phone call follow-up — A nurse will call the patient to counsel patients on their medications and following up with their primary care provider.
  Arms: Follow-up phone call from Nurse
Other: Satisfaction survey — Patients will be given a satisfaction survey.
  Arms: Satisfaction survey
Other: Control group --- no intervention — Control group
  Arms: Control group

SUMMARY:
The investigators hypothesize that the acquisition and correct utilization of medications as well as arranging and attending follow-up appointments will improve as a result of a phone call intervention 1-3 days after elderly patients are discharged from the emergency department (ED).

DETAILED DESCRIPTION:
Older patients seen in the ED are at high risk of functional decline and return visits to the ED. Previous studies have shown that a comprehensive assessment by a geriatric specialist at the time of discharge from the ED along with extensive integration with home services and/or referral to community services can decrease functional decline and return visits to the ED as well as increase patient satisfaction, but this intervention is resource intensive requiring a geriatric discharge specialist to be available to the emergency department 24 hours a day/ 7 days a week. It is also known that in other patient populations telephone reminders to make follow up appointments can increase rate of follow up and that comprehension of discharge instructions is the primary barrier to compliance with discharge instructions. It has been shown that telephone follow-up interviews are feasible for geriatric patients discharged from the ED, and that many elderly patients discharged from the ED do not understand their discharge instructions or attend follow-up appointments. However, there are no published studies evaluating whether a follow up telephone call after discharge from the ED can improve patient compliance with the medical treatment plan including obtaining follow - up appointments and obtaining prescribed medications as well as using them appropriately. We seek to determine if we can increase compliance with medications and outpatient follow up with a phone call from a nurse provider 1-3 days after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or over
* Discharged from the UNC emergency department

Exclusion Criteria:

* In the hospital at the time of phone call follow-up
* Neither the patient nor their responsible party are able to pass a standardized test to assess cognitive function

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 157 (Actual)
Dates: Start 2010-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Whether patient obtained medications prescribed at their discharge from ED | 5-8 days after discharge from ED
Whether patient is using medications that were prescribed at their ED discharge correctly | 5-8 days after discharge from ED
Whether the patient arranged a follow-up appointment with their primary care provider | 5-8 days after discharge from ED
Whether patient attended visit with their primary care provider after discharge from the ED | 30-35 days after discharge from ED

SECONDARY OUTCOMES:
Patient's satisfaction with ED visit | 5-8 days after discharge from the ED
Return to the ED within 30 days of initial visit | 30-35 days after discharge from ED
Cost of the intervention | 35 days after last patient enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Kevin J Biese, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Emergency Department, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Biese K, Lamantia M, Shofer F, McCall B, Roberts E, Stearns SC, Principe S, Kizer JS, Cairns CB, Busby-Whitehead J. A randomized trial exploring the effect of a telephone call follow-up on care plan compliance among older adults discharged home from the emergency department. Acad Emerg Med. 2014 Feb;21(2):188-95. doi: 10.1111/acem.12308. PMID 24673675